CLINICAL TRIAL: NCT01112033
Title: Biliverdin Reductase A in Chronic Hepatitis C Virus Infection
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Military University Hospital, Prague (Other); General University Hospital, Prague (Other); Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Iva Subhanova, Institute of Medical Biochemistry and Laboratory Diagnostics, Charles University, Czech Republic
Other Study IDs: BLVRA1
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C, Chronic
Keywords: biliverdin reductase; BLVRA; hepatitis C; HCV; peripheral blood mononuclear cells; PBMC; liver; genetic polymorphisms
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood, liver biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic HCV infection: The study was performed on therapeutically naïve patients with chronic HCV infection. Patients with positivity of anti-HCV antibodies, and detectable HCV RNA in serum for at least 6 months, were included in the study.

SUMMARY:
In this project, the investigators aim to study the role of biliverdin reductase A (BLVRA) in HCV infected patients prior and during/after standard antiviral therapy in association with viral clearance, disease progression and treatment response and in comparison with healthy subjects.

DETAILED DESCRIPTION:
1. To analyze biliverdin reductase (BLVRA) expression in the liver of HVC infected patients undergoing liver biopsy followed by standard antiviral treatment (peg-interferon plus ribavirin combination therapy) and patients with other forms of liver diseases undergoing liver biopsy as controls.
2. To analyze BLVRA expression in peripheral blood leukocytes (PBL) of therapeutically naïve HCV patients, during/after standard antiviral therapy and healthy controls.
3. To analyze BVLRA genetic polymorphisms both in HCV infected patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

BLVRA expression study

* Therapeutically naïve HCV patients undergoing antiviral treatment with peg-interferon plus ribavirin combination therapy

BLVRA genetic polymorphisms study

* HCV infected patients prior, during, after or without antiviral therapy

Exclusion Criteria:

* Co-infection with HAV, HBV and HIV
* Disorders of heme metabolism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Estimated enrollment: BLVRA expression study: 50 - 100 HCV patients 50 healthy volunteers Polymorphisms of BLVRA study: 300 HCV patients
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To assess differences in BLVRA expression in the liver and PBMC in HCV infected patients in responders and non-responders to standard antiviral therapy. | 72 weeks

SECONDARY OUTCOMES:
To analyze the association of genetic polymorphisms of BLVRA with disease progression and treatment response in HCV infected patients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Iva Subhanova, Principal Investigator — Charles University, Czech Republic
Locations (1):
- Institute of Clinical Biochemistry and Laboratory Diagnostics, First Faculty of Medicine, Charles University in Prague, Prague, Czechia

REFERENCES:
- [Result] Subhanova I, Muchova L, Lenicek M, Vreman HJ, Luksan O, Kubickova K, Kreidlova M, Zima T, Vitek L, Urbanek P. Expression of Biliverdin Reductase A in peripheral blood leukocytes is associated with treatment response in HCV-infected patients. PLoS One. 2013;8(3):e57555. doi: 10.1371/journal.pone.0057555. Epub 2013 Mar 11. PMID 23536765